CLINICAL TRIAL: NCT02048683
Title: A Pharmacokinetic Study of Sevoflurane Inhalation in Burn ICU Patients
Acronym: SEVOBURN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0174; 2013-000960-26
Record Dates: First submitted 2014-01-13; First posted 2014-01-29 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: ICU Patients With Indication of Sedation
Keywords: Pharmacokinetics; Sevoflurane; Burn; Sedation
MeSH Terms: conditions — Burns | interventions — Sevoflurane; Intensive Care Units

ARMS (2):
- burn ICU patients (Experimental): Determination of plasmatic concentrations of sevoflurane at different times of a short term sedation of sevoflurane in burn versus non burn ICU patients
  Interventions: Drug: Short term sedation with sevoflurane in ICU
- non burn ICU patients (Other): Determination of plasmatic concentrations of sevoflurane at different times of a short term sedation of sevoflurane in burn versus non burn ICU patients
  Interventions: Drug: Short term sedation with sevoflurane in ICU

INTERVENTIONS:
Drug: Short term sedation with sevoflurane in ICU

SUMMARY:
Comparing a pharmacokinetic model of a short sevoflurane sedation in burn ICU patients with control ICU patients.

DETAILED DESCRIPTION:
Prospective clinical study in ICU with sedated ventilated patients with sevoflurane with the AnaConda® system, establishing pharmacokinetic model of sevoflurane and its metabolites (hydroxyfluroisopropanol, fluoride) comparing burn and non burn ICU patients

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ventilated requiring invasive procedure in ICU

  * Stable respiratory and hemodynamic conditions
  * Consent of patients or family
  * Arterial line
  * Burn patients : burn area between 20 and 50% (3rd degree) OR non burn patients

Exclusion Criteria:

* BMI <30

  * Sevoflurane anaphylaxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Determination of plasmatic concentrations of sevoflurane | at 5min, 15 min, 60 min and just before the end of sedation.

SECONDARY OUTCOMES:
Determination of plasmatic concentrations of HFIP and fluoride | at 5min, 15 min, 60 min and just before the end of sedation. And 5min, 10 min, 30 min, 60 min and 120 min after the end of sedation

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Perbet S, Bourdeaux D, Lenoire A, Biboulet C, Pereira B, Sadoune M, Plaud B, Launay JM, Bazin JE, Sautou V, Mebazaa A, Houze P, Constantin JM, Legrand M; PRONOBURN group. Sevoflurane for procedural sedation in critically ill patients: A pharmacokinetic comparative study between burn and non-burn patients. Anaesth Crit Care Pain Med. 2018 Dec;37(6):551-556. doi: 10.1016/j.accpm.2018.02.001. Epub 2018 Feb 15. PMID 29455032